CLINICAL TRIAL: NCT00534508
Title: A Study to Determine the Distribution of Tacrolimus in the Skin and the Systemic Pharmacokinetics of Tacrolimus in Adult Patients With Moderate to Severe Atopic Dermatitis Following First and Repeated Application of the Tacrolimus Ointment.
Brief Title: Distribution of Tacrolimus in Skin, Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-30
Record Dates: First submitted 2007-09-21; First posted 2007-09-26 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Dermatitis, Atopic
Keywords: Skin; Pharmacokinetics; Tacrolimus; dermatitis, atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Tacrolimus Ointment 0.1% — Twice daily, 14 days treatment
  Other Names: Protopic 0.1%

SUMMARY:
This study was designed to further increase the understanding of the pharmacokinetics of tacrolimus in the affected skin of atopic dermatitis patients following repeated topical application of tacrolimus ointment 0.1%.

DETAILED DESCRIPTION:
The study was conducted on an out-patient basis, with patients self-administering the ointment twice daily at home. However, on Days 1 and 14 there was only a single application of ointment and this was applied by the Investigator or his/her designee in the clinic. An area of the affected skin was selected for skin biopsy of sufficient size for 5 biopsy samples. The biopsy samples were taken from the same lesion(s) if possible or from an adjacent lesion in the same anatomical area at all times. All areas selected for treatment were treated with tacrolimus ointment 0.1% for a period of two weeks with a follow up period of one week. Two pharmacokinetic profiles (Days 1 and 14) and five skin biopsy samples (Days 1, 2, 15, 18 and 21) were taken.

ELIGIBILITY:
Inclusion Criteria:

* Using the Hanifin and Rajka Criteria, the patient has a diagnosis of moderate to severe atopic dermatitis
* Using the Rajka and Langeland grading system, the patient's atopic dermatitis score is at least 4.5 (moderate to severe)

Exclusion Criteria:

* Patient has a serious skin disorder other than atopic dermatitis.
* Patient has history of eczema herpeticum (defined as an acute disseminated cutaneous herpes simplex type 1 or 2 infection associated with constitutional symptoms like fever, headache, malaise, regional or generalised lymphadenopathy in an individual with eczema).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2000-12; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Distribution of tacrolimus in the skin after first and repeated application of tacrolimus ointment in adult patients with moderate to severe atopic dermatitis. | Days 1, 2, 15. 18 and 21.

SECONDARY OUTCOMES:
Systemic pharmacokinetics of tacrolimus after first and repeated application of tacrolimus ointment in adult patients with moderate to severe atopic dermatitis. | Days 1 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma GmbH
Locations (1):
- Dublin, Ireland

REFERENCES:
- [Background] Undre NA, Moloney FJ, Ahmadi S, Stevenson P, Murphy GM. Skin and systemic pharmacokinetics of tacrolimus following topical application of tacrolimus ointment in adults with moderate to severe atopic dermatitis. Br J Dermatol. 2009 Mar;160(3):665-9. doi: 10.1111/j.1365-2133.2008.08974.x. Epub 2008 Dec 12. PMID 19076975
- [Background] Reitamo S, Mandelin J, Rubins A, Remitz A, Makela M, Cirule K, Rubins S, Zigure S, Ho V, Dickinson J, Undre N. The pharmacokinetics of tacrolimus after first and repeated dosing with 0.03% ointment in infants with atopic dermatitis. Int J Dermatol. 2009 Apr;48(4):348-55. doi: 10.1111/j.1365-4632.2009.03853.x. PMID 19335418